CLINICAL TRIAL: NCT05608148
Title: Clinical Trial of GAIA-102 for Refractory/Relapse Neuroblastomas and Other Malignant Pediatric Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyushu University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAIA-102-PT
Record Dates: First submitted 2022-10-24; First posted 2022-11-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Refractory/Relapse Neuroblastoma; Pediatric Solid Tumors
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GAIA-102 alone (Experimental): GAIA-102: 5 x 10^6 cells / dose at a fixed dose, 1 to 3 doses / week for 3 consecutive weeks
  Interventions: Biological: Biological
- GAIA-102 with Dinutuximab, Filgrastim, Teceleukin combination (Experimental): GAIA-102: 5 x 10^6 cells / dose at a fixed dose, 1 to 3 doses / week for 3 consecutive weeks Filgrastim: 5 µg/kg/day on Day1-14 Teceleukin: 750,000 units/m2/day on Day29-31 and 1,000,000 units/m2/day on Day 36- 39 Dinutuximab: 17.5mg/m2/day on Day4-7 and Day36-39
  Interventions: Biological: Biological
- GAIA-102 with Nivolumab combination (Experimental): GAIA-102: 5 x 10^6 cells / dose at a fixed dose, 3 doses / week for 3 consecutive weeks Nivolumab: 3mg/kg/day(Children) or 240mg/day(Adults) on Day1,15
  Interventions: Biological: Biological
- GAIA-102 with Nivolumab, Teceleukin combination (Experimental): GAIA-102: 5 x 10^6 cells / dose at a fixed dose, 3 doses / week for 3 consecutive weeks Nivolumab: 3mg/kg/day(Children) or 240mg/day(Adults) on Day8,22 Teceleukin: 750,000 units/m2/day on Day1-4 and 1,000,000 units/m2/day on Day 15-18
  Interventions: Biological: Biological

INTERVENTIONS:
Biological: Biological — Intravenous injection of GAIA-102 alone
  Arms: GAIA-102 alone
Biological: Biological — Intravenous injection of GAIA-102 with dinutuximab, filgrastim, teceleukin combination
  Arms: GAIA-102 with Dinutuximab, Filgrastim, Teceleukin combination
Biological: Biological — Intravenous injection of GAIA-102 with nivolumab combination
  Arms: GAIA-102 with Nivolumab combination
Biological: Biological — Intravenous injection of GAIA-102 with nivolumab, teceleukin combination
  Arms: GAIA-102 with Nivolumab, Teceleukin combination

SUMMARY:
Cohort A(GAIA-102 alone):

Confirm the safety of GAIA-102 alone for refractory/relapse neuroblastoma or pediatric solid tumors with lung metastases, and decide recommended dose for Phase II.

Cohort B(GAIA-102 with Dinutuximab):

Confirm the safety of GAIA-102 with Dinutuximab, Filgrastim, Teceleukin combination for refractory/relapse neuroblastoma and decide recommended dose for Phase II.

Cohort C(GAIA-102 with Nivolumab):Confirm the safety of GAIA-102(Follow the recommended doses in Cohort A) with Nivolumab.

Cohort D(GAIA-102 with Nivolumab, Teceleukin):

Confirm the safety of GAIA-102(Follow the recommended doses in Cohort A) with Nivolumab, Teceleukin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been confirmed to have the following malignant tumor by histological examination

   * cohort A : neuroblastoma or malignant solid tumor with pulmonary metastases, rhabdomyosarcoma, undifferentiated sarcoma, Ewing's sarcoma family, osteosarcoma, other cartilage sarcoma, nephroblastoma, hepatoblastoma, germ cell neoplasma, other rare solid tumor (except brain tumor and brain metastases) .
   * cohort B : neuroblastoma.
   * cohort C & D : neuroblastoma and other malignant solid tumors, rhabdomyosarcoma, Ewing's sarcoma family, hepatoblastoma.
2. Undergoing the following treatment.

   * cohort A & B : Patients who have the resistance for more than two treatment regimens, and the resistance for all standard regimens based on the guideline.
   * cohort C & D : Patients with neuroblastoma who have completed the dinutuximab regimen and still have residual tumor. Patients with rhabdomyosarcoma, Ewing's sarcoma family, hepatoblastoma who have the resistance for more than two treatment regimens, and the resistance for all standard regimens based on the guideline.
3. Patients who have medical history for serious side effect , allergy reaction with regards to concomitant drugs.
4. Patients aged from 1years to 24 years at the time of obtaining consent.
5. Patients with performance status(PS) over 50 (Lansky Performance Status Score less than 16 years old) or (Karnofsky Performance Status over 16 years old) at the time of obtaining consent.

Exclusion Criteria:

1. Patients with brain metastases.
2. Patients diagnosed with cancerous meningitis
3. Patients who received allogeneic hematopoietic stem cell transplant.
4. Patients with active autoimmune disease.

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-08-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of Dose Limiting Toxicity(DLT) expression | At the end of Cycle1 (Cohort A & C & D: Cycle period is 28 days, Cohort B: Cycle period is 56 days)
Frequency and severerity of adverse events(Cohort C＆D) | 2 year

SECONDARY OUTCOMES:
Objective reponse rate and presence or absence of new lesions | 2 year
Overall survival rate and progression free survival rate | 2 year
Best overall response and lesion control rate | 2 year
Frequency and severity of adverse events | 2 year
Frequency and severerity of immune-related adverse events | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kyushu University Hospital, Fukuoka, Fukuoka, Japan